CLINICAL TRIAL: NCT00078013
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Examine the Safety and Efficacy of Intravenous MCC-135 as an Adjunct to Standard Therapy With Primary PCI in Patients Diagnosed as Having an ST Elevation Acute Myocardial Infarction
Brief Title: MCC-135 as Adjunct Therapy to Primary Percutaneous Coronary Intervention in ST-Segment Elevation Acute Myocardial Infarction Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCC-135-A02
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Myocardial Infarction
Keywords: AMI; STEMI; Infarct; acute myocardial infarction with ST segment elevation
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Infarction | interventions — MCC 135

INTERVENTIONS:
Drug: MCC-135

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial. The primary objectives of this study are to examine the safety, tolerability, and efficacy of intravenous MCC-135 in limiting final infarct size, as measured by single photon emission computed tomography (SPECT), in patients who require percutaneous coronary intervention (PCI) for a first-documented ST-segment elevation acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Patients will be male or female aged 18 years and older who present to the emergency room (ER) < 6 hours from onset of AMI symptoms. The AMI must be confirmed by a 12-lead electrocardiogram (ECG) and documented in at least 2 leads. Each potential patient must be a candidate for primary PCI and not have thrombolytic therapy planned. To be eligible, patients must not have a prior history of ST-segment elevation MI.

Patients will be randomized in a 1:1:1 ratio to 1 of 3 treatment groups: A, B, and C. Group A will receive MCC-135 4.5 mg/kg/48 hours; Group B will receive MCC-135 9.0 mg/kg/48 hours; and Group C will receive placebo/48 hours. Three hundred thirty patients with a TIMI flow grade of 0/1 are required to complete the study. Because patients will be enrolled and will receive study medication prior to assessment of TIMI flow, it is expected that at least 414 patients may need to be randomized in order to obtain the required 330 qualified patients. All randomized patients will receive 48 hours of study medication, with ongoing assessments during this period, and will have follow-up assessments on Days 3, 4, 5, 30, and 180 as described below, regardless of preoperative TIMI flow grade.

Following initial physical examination, vital signs, establishment of a separate and dedicated IV access, baseline blood sampling, and confirmation of all study eligibility requirements, patients will be randomized and begin receiving study drug as an adjunct to standard therapy. Patients will begin study drug infusion as soon as possible, but < 6 hours following onset of AMI symptoms (i.e., symptoms of myocardial ischemia). Examples of ischemic symptoms include chest, arm, and/or jaw pain, shortness of breath, nausea, diaphoresis, or other symptoms that the investigator considers to be of ischemic origin. A negative result from a urine pregnancy test must be obtained for females of childbearing potential prior to the start of study drug infusion.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent must be obtained from the patient (or, in accordance with state and federal laws and IRB regulations, emergency consent procedures may be employed) before enrollment into the study.
2. The patient is a male or female at least 18 years of age.
3. The patient has an estimated weight between 50 kg (110 lbs) and 140 kg (308 lbs).
4. The patient is suspected to have his/her first-documented ST-segment elevation AMI.
5. The patient has symptoms of ischemia of at least 20 minutes continuous duration, the onset of which occurred < 6 hours prior to study drug infusion. Examples of ischemic symptoms include chest, arm, and/or jaw pain, shortness of breath, nausea, diaphoresis, or other symptoms that the investigator considers to be of ischemic origin.
6. The patient has

   * Anterior MI: > 2 mm ST elevation in at least two contiguous leads out of V1-V4
   * Inferior MI: > 2 mm ST elevation in at least two of II, III, and aVF, with > 10 mm elevation summed for all leads (14, 15)
   * Infero-apical MI: > 1 mm ST elevation in at least two of II, III, and aVF, with both V5 and V6
   * Infero-lateral MI: > 1 mm ST elevation in at least two of II, III, and aVF, with both I and aVL
   * Infero-posterior MI: > 1 mm ST elevation in II, III, and aVF, with > 1 mm ST depression in at least two leads out of V1-V3
7. The patient is expected to undergo primary PCI within 8 hours from the onset of ischemic symptoms (see Inclusion Criterion #5 above).
8. Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria

1. The patient has a past history of ST-segment elevation MI.
2. The patient has a pathologic arrhythmia or is considered electrically unstable (K+, Ca2+).
3. The patient has thrombolytic therapy planned.
4. The patient is in cardiogenic shock unresponsive to IV fluid.
5. The patient has severe bradycardia with heart rate <45 beats/minute.
6. The patient has a pre-existing diagnosis of chronic heart failure (NYHA class III-IV).
7. The patient has left bundle branch block.
8. The patient has any cardiomyopathy or pericarditis.
9. The patient has a history of clinically significant bleeding within the last 3 months.
10. The patient has had any type of major trauma, major surgery, or eye, spinal cord, or brain surgery within the last 3 months that, in the opinion of the investigator, would compromise the patient's response to the standard of care.
11. The patient has a history of clinically significant hepatic disturbance.
12. The patient has a history of chronic renal impairment.
13. The patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the last 6 months.
14. The patient is a woman who is pregnant or lactating.
15. The patient is currently receiving therapy with catecholamines/sympathomimetics, phosphodiesterase inhibitors, or phosphodiesterase inhibitors with calcium sensitizing activity. Patients will be permitted to enter the study if these drugs were discontinued more than 5 half-lives prior to randomization.
16. The patient has a history of multiple drug allergies (including contrast media).
17. The patient has epilepsy or a history of seizures requiring treatment (this does not include febrile seizures as a child).
18. The patient participated in an investigational drug or device study within the last 3 months.
19. The patient has a current dependence on alcohol or history of other drugs of abuse.
20. The patient has current clinically significant psychiatric or neurologic disease or any other condition that, in the investigator's opinion, would prevent adherence to the requirements of the protocol.
21. The patient is clinically significantly immunocompromised (including, but not limited to AIDS and immune-suppressive therapy [i.e., chemotherapy, radiation, systemic corticosteroids]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414
Dates: Start 2003-04; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital/ Harvard Medical School, Boston, Massachusetts, United States